CLINICAL TRIAL: NCT02505438
Title: Application of Deuterated Water (D2O) to Define the Etiology of Musculoskeletal Decline in Ageing and the Efficacy of Nutritional Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DMTD2O13
Record Dates: First submitted 2015-05-08; First posted 2015-07-22 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Young Unilateral Exercise (Experimental): Young Individuals (18-30y) studied before and after 6 weeks unilateral resistance exercise training
  Interventions: Behavioral: Exercise
- Old Unilateral Exercise (Experimental): Old individuals (65-75y) studied before and after 6 weeks of unilateral resistance exercise training
  Interventions: Behavioral: Exercise
- Old Unilateral Exercise and HMB (Experimental): Old individuals (65-75y) studied before and after 6 weeks of unilateral resistance exercise training with HMB (beta-hydroxy-beta-methylbutyrate) supplementation
  Interventions: Behavioral: Exercise
- Old Unilateral Exercise and Omega 3 (Experimental): Old individuals (65-75y) studied before and after 6 weeks of unilateral resistance exercise training with Omega 3 supplementation
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
Maintaining muscle mass and function is important in healthy ageing to maintain quality of life. Loss of muscle mass is major problem, as beyond the age ~50, muscle mass declines by ~1-2% a year. To prevent this loss, the investigators need to understand the mechanism regulating muscle mass as we age. In this project the investigators aim to determine these mechanisms using a new technique of heavy water ingestion, this allows measurement of multiple aspects of skeletal muscle mass metabolism e.g. protein synthesis, over long periods (6 weeks) as people go about their normal everyday activities. The investigators also aim to determine the influence of resistance exercise training on older muscle, as well as differences between men and women in muscle responses to exercise and nutrition HMB (beta-hydroxy-beta-methylbutyrate).

ELIGIBILITY:
Inclusion Criteria:

* Young (18-30y) and old (60-75y) individuals who are generally healthy and recreationally active

Exclusion Criteria:

* Active cardiovascular disease
* Cerebrovascular disease including previous stroke, aneurysm (large vessel or intracranial)
* Respiratory disease including pulmonary hypertension or Chronic obstructive pulmonary disease, Hyper/ hypo parathyroidism, hyper/ hypothyroidism,
* Cushing's disease, diabetes
* Active inflammatory bowel disease
* Renal disease
* Malignancy
* Recent steroid treatment (within 6 mo), or hormone replacement therapy Clotting dysfunction
* Musculoskeletal or neurological disorders
* Any disease requiring long-term drug prescriptions, including statins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | 0-6 Weeks
  Comparison of muscle protein synthesis between young and older individuals and in response to 6 weeks unilateral exercise training and supplementation
Muscle Strength | 0-6 Weeks
  Maximal voluntary contractions of the quadriceps will be performed (leg extension) in the trained and untrained legs. This will be performed at baseline and repeated throughout to monitor training progression

CONTACTS AND LOCATIONS:
Overall Officials: Ken Smith, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital Medical School, Derby, United Kingdom